CLINICAL TRIAL: NCT02606474
Title: Incidence of Placenta Accreta & it's Complications in Cases of Previous Cesarean With Placenta Previa Anterior
Brief Title: Placenta Accreta&Its Complications in Placenta Previa Cases
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Kasr El Aini Hospital (Other)
Responsible Party: Principal Investigator, suzy abdelaziz Abdelhamid, lecturer of obgyn., Kasr El Aini Hospital
Other Study IDs: Obgyn. . .
Record Dates: First submitted 2015-11-07; First posted 2015-11-17 (Estimated); Last update posted 2015-11-17 (Estimated); Status verified 2015-11

CONDITIONS: Placenta Accreta in Placenta Previa Anterior

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
Cases of previous cesarean with placenta previa anterior underwent cesarean section. Placenta accreta is diagnosed during cesarean section &confirmed by pathology. All complications are monitored in cases with placenta accreta and without.

DETAILED DESCRIPTION:
100 cases of gestational age 30 weeks or more with placenta previa anterior with previous one or more cesarean section will be enrolled. History,examination &routine investigations will be taken. Colour doppler will be done to diagnose cases with suspected placenta accreta. Pre & postoperative Hb concentration will be taken. Cases with nonseparation of the placenta will be diagnosed as accreta & confirmed by pathology. Operative time & complications like bladder or intestinal injury will be noted. All data will be analyzed.

ELIGIBILITY:
Inclusion Criteria:

* all pregnant women more than 30 weeks with previous one or more cesarean section with placenta previa anterior

Exclusion Criteria:

* pregnant with unscarred uterus
* scars other than cesarean section

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Pregnant with gestational age more than 30 weeks with previous one or more cesarean section with placenta previa anterior
Sampling Method: Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2015-11; Primary Completion 2016-03 (Estimated); Study Completion 2016-03 (Estimated)

PRIMARY OUTCOMES:
Number of patients with placenta accreta. | 3 months
Number of patients with bladder injury. | 3 months
Number of patients with intestinal injury. | 3 months
Number of patients with cesarean hysterectomy. | 3 months
Number of deaths. | 3 months